CLINICAL TRIAL: NCT00448461
Title: Comparison of Bivalirudin and Unfractioned Heparin in Elective Percutaneous Coronary Interventions
Brief Title: Antithrombotic Regimens and Outcome
Acronym: ARNO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Careggi Hospital (Other)
Responsible Party: David Antoniucci, Division of Cardiology, Careggi Hospital, Florence, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: arcard2007/001
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; percutaneous coronary interventions
MeSH Terms: conditions — Coronary Artery Disease | interventions — Heparin; bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): heparin
  Interventions: Drug: heparin
- 2 (Active Comparator): bivalirudin
  Interventions: Drug: bivalirudin

INTERVENTIONS:
Drug: heparin — comparison between heparin and bivalirudin
  Arms: 1
Drug: bivalirudin — comparison between heparin and bivalirudin
  Arms: 2

SUMMARY:
PROTOCOL SYNOPSIS Title: Comparison of bivalirudin and unfractioned heparin (UFH)+ protamine in elective percutaneous coronary interventions (PCI)

Design: Prospective, randomized, controlled trial

Hypothesis: Bivalirudin is superior to UFH + protamine for the improvement of outcomes in patients undergoing elective PCI

Key Inclusion Criteria:

Patients older than 18 years of age to undergo PCI Clopidogrel loading > 6 hrs prior to PCI according to the PCI guidelines Informed, written consent

Key Exclusion Criteria:

ST-elevation myocardial infarction within the prior 48 hours Active bleeding, bleeding diathesis, recent surgery Severe renal failure Chronic coronary artery occlusion to be treated

Primary endpoint:

Inhospital major bleeding

Secondary endpoints:

1. Composite rate of death, myocardial infarction (MI) or target vessel revascularization (TVR) inhospital, and at 6 months
2. Composite rate of inhospital death, MI or TVR and major bleeding
3. Major and minor bleedings
4. Total vascular complications
5. Post-procedure renal failure

Randomization:

Bivalirudin versus unfractioned heparin followed by protamine at the end of the PCI procedure

Sample size:

Assumed incidence of inhospital major bleeding of 6% in UFH + protamine and of 2% in bivalirudin group; for a power of 80% and a level of 0.05 for each group 425 patients are needed. An interim analysis will be performed after the enrolment of 425 (50%) patients.

Follow-up:

Inhospital, and 6-month clinical follow-up (out-patient clinic or by phone)

DETAILED DESCRIPTION:
Bivalirudin, a direct thrombin inhibitor, has been recently introduced as an alternative to UFH given several important biologic and pharmacokinetic advantages.1,2 In contrast to UFH, it acts independently of antithrombin and inhibits both free and clotbound thrombin; it is not neutralized by circulating inhibitors; does not bind to plasma protein and cause thrombocytopenia.1,2 In the Bivalirudin Angioplasty Study, bivalirudin was associated with a 45% reduction in the relative risk for the composite of death, myocardial infarction, revascularization or hemorrhage as compared to UFH among patients with unstable angina undergoing percutaneous coronary angioplasty.3 Recently, in another randomized trial of patients with intermediate risk undergoing coronary stenting after varying pre-treatment intervals with different doses of thienopyridines, use of bivalirudin was estimated to result in 38% reduction in the relative risk of death, myocardial infarction, urgent repeat revascularization or in-hospital major bleeding at 30 days compared to UFH.4 In addition, bivalirudin was associated with a similar rate of ischemic events and less major bleeding and estimated to be more cost-effective than abciximab administered in adjunct to UFH.4,5 However, previous studies have included patients treated with plain balloon angioplasty or stenting after inadequate pretreatment with thienopyridines (ticlopidine or clopidogrel). Recent guidelines recommend that all patients undergoing PCI must receive a loading dose of 300 - 600 mg of clopidogrel.6 Clopidogrel is a thienopyridine that acts by irreversibly inhibiting the platelet adenosine 5'- diphosphate (ADP) receptor. Compared to ticlopidine, it has the advantage of a more favourable side effect profile 7, 8 and more rapid onset of action.9 Pre-treatment with clopidogrel has been associated with better outcomes among patients undergoing PCI.10-12 After a loading dose of 600 mg, maximum inhibition of aggregation with clopidogrel is achieved within two hours.13 The Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment (ISAR-REACT) trial showed that after pre-treatment with 600 mg clopidogrel for at least 2 hours before intervention, additional use of abicximab to UFH was not associated with any clinically measurable benefit among low-to-intermediate risk patients who underwent PCI.14 On the other hand, patients who received abciximab had a higher rate of thrombocytopenia and more frequently required blood transfusions. Thus, an antithrombotic strategy consisting of a loading dose of 600 mg clopidogrel in addition to UFH and aspirin is a safe and effective way to improve patients' outcomes and reduce costs after PCI. There are few data about the use of protamine neutralization of circulating heparin after successful stent implantation.15-18 However, all the previous studies showed no excess in ischemic complications after stent implantation and subsequent protamine administration, with a strong potential for bleeding complication limitation.

Based on the above-mentioned data it can be said that antithrombotic regimens based on either bivalirudin or UFH intraprocedurally followed by protamine neutralization, are effective strategies to reduce ischemic and hemorrhagic complications in patients with coronary artery disease undergoing PCI. At present, it is not known whether bivalirudin is superior to UFH in patients who have been optimally pre-treated with a loading dose of clopidogrel.

We designed this study to assess whether bivalirudin is superior to unfractioned heparin + protamine in patients undergoing PCI. All patients older than 18 years of age, who require coronary angiography for suspected or established coronary artery disease, but without ST-segment changes, will receive a loading dose of 600 mg clopidogrel at least 2 hours prior to the procedure. Eligible patients who do not meet the exclusion criteria and in whom angiography reveals that revascularization is required and the target lesion(s) is (are) amenable to PCI, will be randomized to receive a bolus of 140 U/kg of heparin or bivalirudin to be administered as an intravenous bolus of 0.75 mg/kg prior to the start of the intervention, followed by infusion of 1.75 mg/kg per hour for the duration of the procedure. All patients will receive aspirin indefinitely and clopidogrel for at least 1 month after PTCA or implantation of bare metal stents and for at least 6 months after implantation of drug-eluting stents; clopidogrel treatment for more than 6 months will be encouraged.19 The primary end point of the study is in-hospital major bleeding. The study is designed to show whether bivalirudin is superior to UFH + protamine with respect to the primary end point.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than age 18 to undergo PCI
2. Pretreatment at least 6 hours before PCI with clopidogrel according to the PCI guidelines.
3. Informed, written consent by the patient or her/his legally-authorized representative for participation in the study.

Exclusion Criteria:

1. Recent ST-elevation myocardial infarction within the last 48 hours.
2. Chronic coronary artery occlusion to be treated
3. Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than one year or that may result in protocol non-compliance.
4. Active bleeding, bleeding diathesis, recent surgery (< 15 days)
5. History of gastrointestinal or genitourinary bleeding within the last 6 weeks
6. Treatment with UFH within 6 hours or low-molecular weight heparin within 8 hours before randomization.
7. Treatment with bivalirudin within 24 hours beforerandomization.
8. Severe uncontrolled hypertension >180/110 mmHg unresponsive to therapy
9. Relevant hematologic deviations: hemoglobin < 100 g/L OR platelet count < 100 x 109 /L.
10. Glomerular filtration rate (GFR) < 30 ml/min or serum creatinine > 30 mg/L or dependence on renal dialysis.
11. Known allergy to the study medications: aspirin, clopidogrel, UFH, bivalirudin; stainless steel; true anaphylaxis after prior exposure to contrast media.
12. Known heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be in-hospital major bleeding. | 30 days

SECONDARY OUTCOMES:
Composite rate of death, myocardial infarction (MI) or urgent | 6 months
target vessel revascularization (TVR) inhospital, and at 6 months | 6 months
Composite rate of inhospital death, MI or TVR and major bleeding | 6 months
Major and minor bleedings | 6 months
Total vascular complications | 6 months
Post-procedure renal failure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Study Director — Division of Cardiology, Careggi Hospital, Florence, Italy
Locations (1):
- Division of Cardiology, Careggi Hospital, Florence, Italy